CLINICAL TRIAL: NCT00991146
Title: An Open-label, Efficacy and Safety Study of Canakinumab (Anti-interleukin-1β Monoclonal Antibody) Administered for 6 Months (24 Weeks) in Japanese Patients With the Following Cryopyrin-associated Periodic Syndromes: Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome, or Neonatal Onset Multisystem Inflammatory Disease, Followed by an Extension Phase to Provide Canakinumab to Study Patients Until it is Approved and Marketed in Japan
Brief Title: Efficacy and Safety Study of Canakinumab Administered for 6 Months (24 Weeks) in Japanese Patients With Cryopyrin-associated Periodic Syndromes Followed by an Extension Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2308
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cryopyrin-associated Periodic Syndromes; Familial Cold Autoinflammatory Syndrome; Muckle-Wells Syndrome; Neonatal Onset Multisystem Inflammatory Disease
Keywords: CAPS; FCAS; MWS; NOMID; cryopyrin-associated periodic syndromes; Familial Cold Autoinflammatory Syndrome; Muckle-Wells Syndrome; Neonatal Onset Multisystem Inflammatory Disease; canakinumab; ACZ885; children; systemic autoinflammatory disease; NALP-3; human monoclonal anti-human interleukin-1beta (IL-1beta)antibody; autosomal dominant; familial autoinflammatory syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — canakinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- canakinumab (Experimental)
  Interventions: Drug: canakinumab

INTERVENTIONS:
Drug: canakinumab — canakinumab

SUMMARY:
To date there are no approved effective therapies for the treatment of cryopyrin-associated periodic syndromes (CAPS) including Familial Cold Autoinflammatory Syndrome (FCAS), Muckle-Wells Syndrome (MWS), or Neonatal Onset Multisystem Inflammatory Disease (NOMID) in Japan.

The study will assess the efficacy and safety of canakinumab in Japanese patients with cryopyrin-associated periodic syndromes (CAPS). In previous and currently ongoing CAPS studies (CACZ885A2102, CACZ885D2201, CACZ885D2304, CACZ885D2306), it has been observed that treatment with canakinumab in patients with CAPS contributed to ensure absence of relapse, to improve signs and symptoms and to prevent secondary disease complications. However, no Japanese patients have been included in those studies. This study will allow access for Japanese patients to a new potentially efficacious treatment for CAPS patients with a convenient dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. At study entry, patients should have a clinical diagnosis of FCAS, MWS or NOMID and require medication. At the time of screening, patients can be either untreated or treated with other medication.
2. Presence, or history of at least 2 of the following symptoms:

   * For NOMID patients:

     * Typical NOMID urticarial rash
     * Signs of central nervous system (CNS) involvement such as increased intracranial pressure and/or papilledema and/or cerebral spinal fluid pleiocytosis and/or stroke and/or seizures, and/or sensorineural hearing loss
     * Typical arthropatic changes on X-rays: epiphysal and/or patellar overgrowth With start of NOMID symptoms before or at 6 months of age
   * For MWS patients:

     * periodic fever
     * headache/migraine
     * arthralgia
     * urticarial skin rash
     * conjunctivitis
     * myalgia
     * sensorineural hearing impairment
   * For FCAS patients:

     * urticarial skin rash
     * fever/chills
     * conjunctivitis
     * joint pain
3. Patients requiring oral steroids, NSAIDs and/or disease-modifying antirheumatic drugs (DMARDs) can be enrolled if they are on a stable dose (oral steroids: < 20 mg/day or < or = 0.4 mg/kg prednisone or prednisone equivalent, whichever applies) for at least 4 weeks prior to the screening visit.
4. Able to communicate with the investigator and comply with the requirements of the study (for children the parent can assist when necessary).

Exclusion Criteria:

1. Pregnant or nursing (lactating) women.
2. All women capable of becoming pregnant unless they are postmenopausal or are using one or more methods of contraception.
3. Participation in any other study within 30 days
4. Infection with HIV, Hepatitis B or C.
5. Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose.
6. History of drug or alcohol abuse within the 12 months prior to dosing.
7. Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing for adults.
8. History of significant medical conditions, which in the doctor's opinion would exclude the patient from participating in this trial.
9. History of renal transplantation.
10. Presence of any additional rheumatic diseases or significant systemic diseases. For example, major chronic infectious/ inflammatory/ immunologic disease (such as inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, systemic lupus erythematosus in addition to the autoinflammatory disease).
11. Presence of any of the following laboratory abnormalities: ALT or AST greater than 2 times the upper limit of normal (ULN), platelet count less than 100x109/L.
12. History of recurrent and/or evidence of clinically significant active bacterial, fungal, or viral infections.
13. History of contact with patients with suspected tuberculosis symptoms; or history or complication of tuberculosis infection.
14. Use of the following therapies:

    * Etanercept in the 4 weeks prior to the baseline visit (Day 1) and thereafter
    * Adalimumab in the 8 weeks prior to the baseline visit (Day 1) and thereafter
    * Infliximab in the 12 weeks prior to the baseline visit (Day 1) and thereafter
    * Rituximab in the 26 weeks prior to the baseline visit (Day 1) and thereafter
    * Tocilizumab in the 3 weeks prior to the baseline visit (Day 1) and thereafter
    * Any other investigational biologics in the 8 weeks prior to the baseline visit (Day 1) and thereafter (with the exception of anakinra therapy-see below)
    * Anakinra therapy after the baseline visit (Day 1). Last anakinra injection should occur not less than 6 hours prior to the canakinumab injection at Day 1
    * Leflunomide in the 4 weeks prior to the baseline visit (Day 1) and thereafter. After the completion of leflunomide treatment a cholestiramine in dose 8 g 3 times per day for 14 days is recommended.
    * Thalidomide in the 4 weeks prior to the baseline visit (Day 1) and thereafter
    * Cyclosporine in the 4 weeks prior to the baseline visit (Day 1) and thereafter
    * i.v. immunoglobulin (i.v. Ig) in the 8 weeks prior to the baseline visit (Day 1) and thereafter
    * 6-Mercaptopurine, azathioprine, cyclophosphamide, or chlorambucil in the 12 weeks prior to the baseline visit (Day 1) and thereafter
    * Dapsone, mycophenolate mofetil in the 3 weeks prior to the baseline visit (Day 1) and thereafter
    * > or = 20 mg/day or >0.4 mg/kg, whichever applies, of prednisone or prednisone equivalent in the 4 week prior to the baseline visit (Day 1) and thereafter
    * Methyl prednisone pulse therapy in the 4 weeks prior to baseline visit and thereafter
15. History of allergic reaction to similar drugs. No additional exclusions may be applied by the doctor, in order to ensure that the study population will be representative of all eligible patients.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of participants without a relapse | 24 weeks

SECONDARY OUTCOMES:
Number of complete responder patients | 29 days
Clinical improvement (or resolution) with regards to: central nervous system (CNS) involvement, eye disease, hearing impairment, skin disease, joint disease, fever, and kidney function | 24 months
Number of patients experiencing a relapse during the entire study | 24 months
How much canakinumab is contained in the patients' blood (pharmacokinetics) and what are the effect of canakinumab on the patients' body (pharmacodynamic) | 24 months
Presence of antibody against canakinumab | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto

REFERENCES:
- [Result] Imagawa T, Nishikomori R, Takada H, Takeshita S, Patel N, Kim D, Lheritier K, Heike T, Hara T, Yokota S. Safety and efficacy of canakinumab in Japanese patients with phenotypes of cryopyrin-associated periodic syndrome as established in the first open-label, phase-3 pivotal study (24-week results). Clin Exp Rheumatol. 2013 Mar-Apr;31(2):302-9. Epub 2013 Feb 1. PMID 23380020